CLINICAL TRIAL: NCT06246370
Title: Kronik Obstruktif Akciğer Hastalığında Servikal bölge Biyomekaniği, Kas Performansı ve Solunum Kas Kuvvetinin İncelenmesi
Brief Title: An Investigation of the Cervical Region Biomechanics in Patients With Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, PT, PhD, Assoc. Prof., Hacettepe University
Other Study IDs: GO 23/616
Record Dates: First submitted 2023-10-11; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Postural; Defect; Cervical Pain; Cough
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Neck Pain; Cough

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD group: patients with COPD aged 40 years and above.
- control group: aged matced healty patients

SUMMARY:
The aim of this study is to investigate cervical region biomechanics, muscle performance and respiratory muscle strength in patients with Chronic Obstructive Pulmonary Disease (COPD) compared to healthy subjects.

DETAILED DESCRIPTION:
The secondary purposes are to investigate the correlation between cervical region biomechanics and posture, functional exercise capacity, depression &anxiety level,neck disability, cough severity. In accordance with this purposes, 17 patients with COPD who have Global Initiative for Chronic Obstruction Lung Disease (GOLD) stage 1-2-3-4, being clinically stable for 4 weeks and 17 healthy controls will be included ages>40. Tests and questionnaires will be used in order to determine the severity of COPD and to evaluate posture. Photographical analysis in lateral and posterior views will be used for evaluation of cranioservical region static and dynamic biomechanics. To analyze of chest wall, radiographic evaluation will be performed. Goniometry will be used for evaluation dynamic craniocervical kinematic analysis. Cranioservical region muscle strength and endurance tests will be performed. Respiratory muscle strength tests and cough evaluation test will be performed. Neck disability index, cough evaluation test questionnare, beck depression and anxiety questionnares, Nordic Musculoskeletal questionnare will be used. 6 Minute Pegboard and Ring Test, 6 Minute Walk Test will be performed. According to the results to be obtained, relationship between cranioservical region biomechanics and posture will be investigated based on the severity of disease in patients with COPD. It will guide professional working in the field.

ELIGIBILITY:
Inclusion Criteria:

* • Being diagnosed with stage 1-2-3-4 according to the Classification of Airflow Limitation in COPD (GOLD) system,

  * Being >40 years old,
  * Being cognitively competent to understand and answer evaluation questions.
  * Being clinically stable for the last 4 weeks,
  * Being under control of accompanying comorbid conditions (such as hypertension, diabetes),
  * Volunteering to participate in the research.

Exclusion Criteria:

* • Having been hospitalized due to exacerbation in the last 3 months,

  * Having a musculoskeletal, neurological, rheumatological or oncological disease that affects the craniocervical & cervicothoracic joints and/or may prevent evaluation,
  * Having undergone any surgical intervention on the craniocervicofacial region and spine in the last six months,
  * Having lung malignancy, neoplasm, adenocarcinoma,
  * Being a lung cancer patient or having received cancer treatment (head and neck lung radiotherapy), having undergone pneumonectemia, lobectomy or resection surgery,
  * Being treated for anxiety and depression,
  * Having scoliosis,
  * Having a congenital anomaly of the craniocervicofacial region.
  * Having 3 out of 4 findings according to the diagnostic criteria for cervical radiculopathy,
  * Having thoracic outlet syndrome (TOS)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred by the department of chest diseases of Hacettepe university will be taken
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2024-09-06 (Estimated); Study Completion 2025-09-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of sagittal cobb angle | day 1
  Cobb anle will measure from X-ray imagination between T2- T12 level.
Cranial rotation angle | day 1
  Tragus- eye horizontal angle will measure from lateral cervical photographs.
evaluation of cervical region biomechanic (dynamic) | day 1
  Investigation of the cervical region range of motions of cervical flexion, cervical extension, cervical lateral flexion, and cervical rotation range of motion.
cervical inclination angle | day 1
  tragus eye and C7 level horizontal angle will measure from lateral cervical photographs.
cervical lateral flexion angle | day 1
  the angle between pogonion-tragus and C7 level will measure from lateral cervical photographs.
Shoulder elevation/depression angle | day 1
  the angle between acromion- C7 level and horizontal line will measure from lateral cervical photographs.
chest wall analysis | day 1
  the distance between 3rd, 7th and 9th ribs and horizontal line will measure from X-Ray
rib angle | day 1
  Sternum and 4th,5th, 6th rib will mark and the angle between these and maximum anteroposteror dimention of the thorax will measure from X-Ray.
diaphragma height | day 1
  the distance between T1- and L2 level will measure from X-Ray.

SECONDARY OUTCOMES:
postural analysis | day 1
  investigation of posture by photographic analysis in patients with COPD upward rotation/ anterior tilt/internal rotation of scapula, scapular elevation, and scapular abduction evaluations will measure from photographic analysis.
respiratory muscle strength | day 1
  respiratory muscle strength by mouth pressure device, mean inspiratory pressure and mean expiratory pressure will be tested.
cervical region muscle strength and endurance | day 1
  investigation of cervical region muscle strength and endurance with stabilizer biofeedback pressure method
airway flow limitation | day 1
  severity of disease by Global İnitiative for Chronic Obstructive Pulmonary Disease scale, GOLD 1: FEV1 (predicted%) ≥%80 GOLD 2: %50 ≤ FEV1 (predicted% ) < %79 GOLD 3: %30 ≤ FEV1 (predicted%) < %49 GOLD 4 : FEV1 (predicted%) < %30
management of cough | day 1
  cough severity will be tested by the Cough evaluation Test.(1-5 scaling of items, 5-25 score range) The minimal important difference was 2.
Upper Extremity Functional Capacity | day 1
  evaluation of upper extremity functional capacity with 6-minute pegboard ring test
functional exercise capacity | day 1
  functional exercise capacity by 6 minute walking test.
anxiety level | day 1
  investigation of anxiety level with the Beck Anxiety Questionnaire (A total score of 0-7 is considered minimal range, 8-15 is mild, 16-25 is moderate, and 26-63 is severe)
general musculoskeletal pain level | day 1
  general musculoskeletal pain level is evaluated by Nordic Musculoskeletal Questionnare, cut off point is 'one yes answer'
evaluation of cervical radiculopathy | day 1
  1. Spurling test
  2. cervical distraction test
  3. cervical rotation test (if + spurling and cervical distraction test side is same with this test and is lower than 60 degree)
  4. upper extremity stretching test
  If there are 3 positive answer to 4 tests, cervical radiculopathy existence will be detected.
investigation of neck disability severity | day 1
  evaluation of neck disability level by neck disability index,10-point change should be used as the minimum clinically important difference for patients with upper extremity referred sypmtoms
investigation of the disease severity | day 1
  evaluation of the disease severity with chronic obstructive pulmonary disease severity with Chronic Respiratory Questionnaire MCID( minimal clinically important difference) = a change of 0.5 per item A change in the score of 0.5 on the 7 point scale reflects a clinically significant small change
  A change of 1.0 reflects a moderate change
  A difference of 1.5 represents a large change
investigation of the Pulmonary Function | day 1
  evaluation of pulmonary functions with Lung function test FEV %,FEV1 %, FVC %, FEV1/FVC % , FEF 25-75%, PEF %
cough sufficiency in patients with COPD | day 1
  evaluation of cough sufficiency with peak expiratory flow meter device, A peak expiratory flow of < 80% predicted was the best cut-off to detect airflow limitation.
depression level | day 1
  investigation of depression level with Beck Depression Inventory (cut off point is 17 point) Conventional cutoffs are 0-9 for normal range, 10-18 for mild to moderate depression, 19-29 for moderate to severe depression, and 30-63 for severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Demirel, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Health Sciences Faculty, Ankara, Turkey (Türkiye)